CLINICAL TRIAL: NCT04413773
Title: Use of Simple Explanation Videos to Reduce Perioperative Patient Anxiety in Children.
Brief Title: Patient Anxiety Reduction in Children by Using Simple Explanation Videos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Dr. med. Julian Trah, Medical Doctor, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VideoAnx2020
Record Dates: First submitted 2020-05-27; First posted 2020-06-04 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Perioperative Anxiety
Keywords: Anxiety, Video education, perioperative
MeSH Terms: conditions — Anxiety Disorders | interventions — Therapeutics; Videotape Recording

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (Active Comparator): Treatment as Usual, Explanation of standard procedures before, during and after surgery by nurse
  Interventions: Other: Treatment as usual
- Treatment as usual + Video (Experimental): Treatment as usual and additionally Video
  Interventions: Other: Treatment as usual + Video

INTERVENTIONS:
Other: Treatment as usual + Video — Additionally to treatment as usual a video is shown to participant about procedures on the ward before, during and after surgery
  Arms: Treatment as usual + Video
Other: Treatment as usual — Explanation of standard procedures before, during and after surgery by nurse
  Arms: Treatment as usual

SUMMARY:
The reduction of preoperative anxiety in children and adolescents before an elective surgical procedure is an important clinical question in perioperative care. Adequate, age-appropriate patient information about the processes of the inpatient stay plays an important role in order to address possible worries and fears to reduce.

The medium video is popular with children and adolescents today and offers the possibility of an easily understandable and vivid presentation of information.

DETAILED DESCRIPTION:
Studies by the health insurance companies, scientific publications and economic papers show that in times of increasing economic interests of the hospitals and the resulting necessity of economic working methods in the medical system, less time remains for human interaction. This creates areas of conflict, such as the patient's right to information regarding the time available to medical personnel. This in turn leads to significant stress factors in patients who are involved in the treatment and mostly on the communication level, such as "Missing information", "misunderstood visit", "missing partnership relationship" refer to what is reflected in patient satisfaction and fears. Studies show how important good perioperative psychosocial care is for reducing these circumstances in children, also and especially in the context of further development. The drug options for calming and reducing anxiety are already known, but there are also increasing numbers of non-drug approaches to reducing anxiety and stress in the literature. Painting therapy and clinic clowns are examples. However, access to such resources is limited and costs are permanently high. New technologies, e.g. mobile phones and tablets, with the associated media, increasingly finding their way into our society, are now inexpensive to buy and have become an integral part of most households. Such devices and media are increasingly used in clinical studies and patient care. Their use is tested extensively in modern medicine, e.g. to avoid unnecessary postoperative consultations in the emergency room or to increase cognitive learning for children. Even small children can use and understand these media early on. Videos are one of the most common media already understood by the smallest patients.

ELIGIBILITY:
Inclusion Criteria:

1. All patients (children) who present themselves planned in the Altona Children's Hospital or in the University Clinic Hamburg Eppendorf in the course of an upcoming elective operation.
2. The surgical intervention must take place in one of the following body regions: thorax, abdomen and / or extremities (incl. Head and neck)
3. A signed declaration of consent from the parents or legal guardians is available
4. The patient has given a declaration of consent
5. No mental illnesses may be diagnosed
6. No chronic pre-existing conditions may be diagnosed
7. Age of the patients is between 6 and 17 years

Exclusion Criteria:

1. No signed declaration of consent from the parents or legal guardians available
2. There is no signed declaration of consent from the patient

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Change in perioperative Anxiety in Children (T1 vs. T2, TAU vs. Video) | Through study completion, an average of 1 year
  The primary endpoint was to analyze the preoperative state-anxiety in children before (t1) and after (t2) the intervention (video), compared with standard care (TAU). we use State-Trait-Anxiety-Operation-Inventory

SECONDARY OUTCOMES:
Change in perioperative Anxiety in Parental Report (T1 vs. T2, TAU vs. Video) | Through study completion, an average of 1 year
  Secondary endpoint was to analyze the preoperative trait-anxiety in children, as well as the preoperative state- and trait-anxiety in the parental report. We use the State-Trait-Anxiety-Operation-Inventory
Nurse reported anxiety before and after Intervention (T1 vs. T2) | Through study completion, an average of 1 year
  we analyzed the nurse-reported anxiety status of the child before (t1) and after (t2) the intervention, we use a short State-Anxiety-Inventory (Krohne et al. 2005)
Perioperative Anxiety separated in state and trait anxiety (T1 vs T2, TAU vs Video) | Through study completion, an average of 1 year
  difference between anxiety levels, again separated in state and trait, reported by children, We use the State-Trait-Anxiety-Operation-Inventory
Evaluation of STOA in a pediatric cohort | Through study completion, an average of 1 year
  Evaluation of Questionnaire in a pediatric cohort

CONTACTS AND LOCATIONS:
Overall Officials: Julian Trah, MD, Principal Investigator — Department of pediatric surgery
Locations (2):
- Germany (2):
  - University Hospital Hamburg Eppendorf - Department of pediatric surgery, Hamburg
  - The Altona Children's Hospital, Hamburg